CLINICAL TRIAL: NCT03304509
Title: Comparative Study Between Conventional and Telematic Follow-up of Patient Treated in a General Ang GI Surgery Department (TLM-CGD)
Brief Title: Comparative Study Between Conventional and Telematic Patients Follow-up
Acronym: TLM-CGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Manel Cremades, MD, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GermansTIPH
Record Dates: First submitted 2017-09-30; First posted 2017-10-09 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Telemedicine; General Surgery; Outpatients

STUDY DESIGN:
Intervention Model Description: Patients will be included and assigned randomly, using an informatic program, to one of the study arms before hospital discharge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-face follow-up (No Intervention): Face-to-face follow-up after hospital discharge
- Telematic follow-up (Experimental): Telematic follow-up after hospital discharge
  Interventions: Other: Telematic follow-up

INTERVENTIONS:
Other: Telematic follow-up — Telematic follow-up by using a platform with videoconference
  Arms: Telematic follow-up

SUMMARY:
This is a parallel group clinical trial comparing two types of follow-up in patients operated and treated in a General and GI surgery department. Face-to-face vs telematic follow-up by using a platform that offers videoconferencing will be compared.

Patients will be included and assigned randomly to each group using an informatics program until 100 patients are reached in each arm of the study ("n" total = 200 patients) The main and secondary outcomes will be evaluated 30 days after the date of the follow-up.

DETAILED DESCRIPTION:
This is a parallel group clinical trial comparing two types of follow-up in patients operated and treated in a General and GI surgery department. Face-to-face vs telematic follow-up by using a platform that offers videoconferencing will be compared.

The hypothesis is that a follow-up based on a telematic visit will no add extra comorbidities while could reduce costs and increase patients satisfaction.

Patients will be included and assigned randomly to each group using an informatics program until 100 patients are reached in each arm of the study ("n" total = 200 patients) Information regarding the type of follow-up and the instructions to perform the telematic visit will be provided to patients before discharge. The follow-up date will be set according to the established protocol for each type of pathology.

In case of clinical complications patients will be referred to the emergency department or will be visited in face-to-face basis.

The main and secondary outcomes will be evaluated 30 days after the date of the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated or operated in the General and GI Surgery department in "Hospital Germans Trias i Pujol"

Exclusion Criteria:

* Proctological Surgery
* Personal conditions that not allow a correct comprehension or developement of the study
* Patients with postoperative complications greater than Clavien-Dindo grade II
* Not being in possession of the necessary informatic devices in case of telematic follow-up
* Not having a basic informatic knowledge in case of telematic follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-03-19 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Follow-up accomplishment | From date of discharge until the date of follow-up, 30 days after discharge
  Percentage of patients that can finish the follow-up in the assigned group

SECONDARY OUTCOMES:
Emergency department consultation | From discharge until 30 days after the follow-up date
  Comparison between number of emergency department consultations in each group if related to the surgical procedure
Patient satisfaction | 30 days after the follow-up date
  Assessment of the patient satisfaction related to the follow-up using the NHS Outpatients Questionnaire. The results will be the comparision of percentage of each answer in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Manel Cremades, MD, Principal Investigator — General and GI Surgical Department Staff
Locations (1):
- Hospital Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
All the study will be carried out in our institution and no individual data will be shared with other researchers or investigation centers unless if needed to support our study results

REFERENCES:
- [Background] Johnston MJ, King D, Arora S, Behar N, Athanasiou T, Sevdalis N, Darzi A. Smartphones let surgeons know WhatsApp: an analysis of communication in emergency surgical teams. Am J Surg. 2015 Jan;209(1):45-51. doi: 10.1016/j.amjsurg.2014.08.030. Epub 2014 Oct 22. PMID 25454952
- [Background] Khanna V, Sambandam SN, Gul A, Mounasamy V. "WhatsApp"ening in orthopedic care: a concise report from a 300-bedded tertiary care teaching center. Eur J Orthop Surg Traumatol. 2015 Jul;25(5):821-6. doi: 10.1007/s00590-015-1600-y. Epub 2015 Jan 30. PMID 25633127
- [Background] Kvedar J, Coye MJ, Everett W. Connected health: a review of technologies and strategies to improve patient care with telemedicine and telehealth. Health Aff (Millwood). 2014 Feb;33(2):194-9. doi: 10.1377/hlthaff.2013.0992. PMID 24493760
- [Background] Armstrong KA, Coyte PC, Bhatia RS, Semple JL. The effect of mobile app home monitoring on number of in-person visits following ambulatory surgery: protocol for a randomized controlled trial. JMIR Res Protoc. 2015 Jun 3;4(2):e65. doi: 10.2196/resprot.4352. PMID 26040252
- [Background] Dobke MK, Bhavsar D, Gosman A, De Neve J, De Neve B. Pilot trial of telemedicine as a decision aid for patients with chronic wounds. Telemed J E Health. 2008 Apr;14(3):245-9. doi: 10.1089/tmj.2007.0038. PMID 18570547
- [Background] Weinstein RS, Lopez AM, Joseph BA, Erps KA, Holcomb M, Barker GP, Krupinski EA. Telemedicine, telehealth, and mobile health applications that work: opportunities and barriers. Am J Med. 2014 Mar;127(3):183-7. doi: 10.1016/j.amjmed.2013.09.032. Epub 2013 Oct 29. PMID 24384059
- [Background] Shah MN, Wasserman EB, Gillespie SM, Wood NE, Wang H, Noyes K, Nelson D, Dozier A, McConnochie KM. High-Intensity Telemedicine Decreases Emergency Department Use for Ambulatory Care Sensitive Conditions by Older Adult Senior Living Community Residents. J Am Med Dir Assoc. 2015 Dec;16(12):1077-81. doi: 10.1016/j.jamda.2015.07.009. Epub 2015 Aug 17. PMID 26293419
- [Background] Eisenberg D, Hwa K, Wren SM. Telephone follow-up by a midlevel provider after laparoscopic inguinal hernia repair instead of face-to-face clinic visit. JSLS. 2015 Jan-Mar;19(1):e2014.00205. doi: 10.4293/JSLS.2014.00205. PMID 25848178
- [Background] Charles BL. Telemedicine can lower costs and improve access. Healthc Financ Manage. 2000 Apr;54(4):66-9. PMID 10915354
- [Background] Pericas JM, Aibar J, Soler N, Lopez-Soto A, Sanclemente-Anso C, Bosch X. Should alternatives to conventional hospitalisation be promoted in an era of financial constraint? Eur J Clin Invest. 2013 Jun;43(6):602-15. doi: 10.1111/eci.12087. Epub 2013 Apr 17. PMID 23590593
- [Background] Bator EX, Gleason JM, Lorenzo AJ, Kanaroglou N, Farhat WA, Bagli DJ, Koyle MA. The burden of attending a pediatric surgical clinic and family preferences toward telemedicine. J Pediatr Surg. 2015 Oct;50(10):1776-82. doi: 10.1016/j.jpedsurg.2015.06.005. Epub 2015 Jun 20. PMID 26195452
- [Background] Rasmussen BS, Froekjaer J, Bjerregaard MR, Lauritsen J, Hangaard J, Henriksen CW, Halekoh U, Yderstraede KB. A Randomized Controlled Trial Comparing Telemedical and Standard Outpatient Monitoring of Diabetic Foot Ulcers. Diabetes Care. 2015 Sep;38(9):1723-9. doi: 10.2337/dc15-0332. Epub 2015 Jun 26. PMID 26116717
- [Background] Sathiyakumar V, Apfeld JC, Obremskey WT, Thakore RV, Sethi MK. Prospective randomized controlled trial using telemedicine for follow-ups in an orthopedic trauma population: a pilot study. J Orthop Trauma. 2015 Mar;29(3):e139-45. doi: 10.1097/BOT.0000000000000189. PMID 24983434
- [Background] Sharareh B, Schwarzkopf R. Effectiveness of telemedical applications in postoperative follow-up after total joint arthroplasty. J Arthroplasty. 2014 May;29(5):918-922.e1. doi: 10.1016/j.arth.2013.09.019. Epub 2013 Dec 15. PMID 24342278
- [Background] Piqueras M, Marco E, Coll M, Escalada F, Ballester A, Cinca C, Belmonte R, Muniesa JM. Effectiveness of an interactive virtual telerehabilitation system in patients after total knee arthoplasty: a randomized controlled trial. J Rehabil Med. 2013 Apr;45(4):392-6. doi: 10.2340/16501977-1119. PMID 23474735
- [Background] Robaldo A, Rousas N, Pane B, Spinella G, Palombo D. Telemedicine in vascular surgery: clinical experience in a single centre. J Telemed Telecare. 2010;16(7):374-7. doi: 10.1258/jtt.2010.091011. Epub 2010 Aug 2. PMID 20679407
- [Background] Fallaize RC, Tinline-Purvis C, Dixon AR, Pullyblank AM. Telephone follow-up following office anorectal surgery. Ann R Coll Surg Engl. 2008 Sep;90(6):464-6. doi: 10.1308/003588408X300975. Epub 2008 Jul 2. PMID 18598594
- [Background] Haukipuro K, Ohinmaa A, Winblad I, Linden T, Vuolio S. The feasibility of telemedicine for orthopaedic outpatient clinics--a randomized controlled trial. J Telemed Telecare. 2000;6(4):193-8. doi: 10.1258/1357633001935347. PMID 11027118
- [Background] Wallace P, Haines A, Harrison R, Barber J, Thompson S, Jacklin P, Roberts J, Lewis L, Wainwright P; Virtual Outreach Project Group. Joint teleconsultations (virtual outreach) versus standard outpatient appointments for patients referred by their general practitioner for a specialist opinion: a randomised trial. Lancet. 2002 Jun 8;359(9322):1961-8. doi: 10.1016/s0140-6736(02)08828-1. PMID 12076550